CLINICAL TRIAL: NCT05073978
Title: The Association Between Niacin Deficiency and Birth Defects: a Case-control Study
Brief Title: B-vitamin Levels and Adverse Pregnancy Outcomes
Status: Completed | Type: Observational
Sponsor: Westlake University (Other)
Collaborators: Beijing Obstetrics and Gynecology Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20210119SHJ001
Record Dates: First submitted 2021-09-22; First posted 2021-10-12 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Birth Defect; Pregnancy Loss; Pregnancy Complications; Pregnancy Induced Hypertension; Recurrent Pregnancy Loss; Health Problems in Pregnancy; Gestational Diabetes; Gestational Hypertension; Preterm Birth
Keywords: vitamin B; pregnancy outcome
MeSH Terms: conditions — Congenital Abnormalities; Pregnancy Complications; Hypertension, Pregnancy-Induced; Diabetes, Gestational; Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — first-trimester maternal blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: Case group with certain pregnancy outcome, e.g., miscarriage, stillbirth, preterm birth, and birth defects,gestational hypertension, gestational diabetes mellitus, etc.
  Interventions: Other: No intervention
- Control group: Control group without certain pregnancy outcome,e.g., miscarriage, stillbirth, preterm birth, and birth defects,gestational hypertension, gestational diabetes mellitus, etc.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study without any intervention

SUMMARY:
This prospective nested case-control study aims to examine the effects of blood vitamin B levels in first-trimester pregnant women on the pregnancy outcomes

DETAILED DESCRIPTION:
Folate deficiency can cause severe adverse pregnancy outcomes, such as neural tube defects. Effective folate functioning requires essential metabolic interactions with other B vitamins including vitamin B2, vitamin B3, vitamin B6, and vitamin B12, which can also influence pregnancy outcomes independently. For example, animal and family studies have identified that niacin (B3) deficiency can lead to congenital malformations. However, how folate and related B-vitamin levels interact with each other while affecting various pregnancy outcomes including abortion, birth defects, pregnancy complications, etc. is unclear. Besides, folate levels in previous studies were mostly measured in plasma which are easily influenced by dietary factors, instead of red blood cell folate which can reflect the long-term status. Moreover, the difference in the risk of neural tube defects across a range of maternal red blood cell folate concentrations has been largely ignored. Using data of pregnant women recruited at Beijing Obstetrics and Gynecology Hospital from December 2020 to December 2021, this case-control study aims to examine the association of folate and related B-vitamin levels in first-trimester blood samples (plasma and red blood cell) with pregnancy outcomes, particularly the association between niacin deficiency and birth defects.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with 6-13(+6 days) gestational weeks
* Resided in Beijing in the past year
* Pregnant women who intend to have antenatal examinations and delivery at Beijing Obstetrics and Gynecology Hospital
* Pregnant women who are willing to participate in this study with informed consent

Exclusion Criteria:

* Women with Hepatitis B, syphilis, HIV/AIDS and other infectious diseases.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: all pregnant women recruited in the birth cohort of Beijing Obstetrics and Gynecology Hospital between 2020.12 to 2021.12
Sampling Method: Non-Probability Sample
Enrollment: 7500 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
fetal outcomes | at delivery
  Including intrauterine growth retardation,abortion, stillbirth, preterm birth, live birth
fetal outcomes | 42 days after delivery
  Including birth defects
maternal outcomes | at delivery
  Including gestational hypertension, preeclampsia, gestational diabetes mellitus, hypothyroidism

CONTACTS AND LOCATIONS:
Overall Officials: Hongjun Shi, PhD, Principal Investigator — Westlake University
Locations (1):
- Beijing Obstetrics and Gynecology Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided